CLINICAL TRIAL: NCT04598854
Title: The Investigation of Therapeutic Effect and Molecular Mechanism After Intravascular Laser Irradiation of Blood for Osteoarthritis of Knee
Brief Title: Intravascular Laser Irradiation of Blood for Osteoarthritis of Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Liang-Cheng Chen, Clinical Professor of Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 109WFE0110237
Record Dates: First submitted 2020-10-18; First posted 2020-10-22 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-03

CONDITIONS: Osteoarthritis, Knee
Keywords: Intravascular laser irradiation of blood; Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: The treatment group will receive an intravenous helium-neon laser phototherapy. A vein indwelling needle will be placed in their veins located in the upper elbow, and the laser fiber catheter will be introduced through the indwelling cannula. The power is set between 2.5 ~ 3.0Mw, 60 minutes each time, once a day for five consecutive days. The steps for the control group are the same, except that the output power is adjusted to zero intensity.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): The treatment groupreceive an intravenous helium-neon laser phototherapy. A vein indwelling needle will be placed in their veins located in the upper elbow, and the laser fiber catheter will be introduced through the indwelling cannula. The power is set between 2.5 ~ 3.0Mw, 60 minutes each time, once a day for five consecutive days. The steps for the control group are the same, except that the output power is adjusted to zero intensity.
  Interventions: Device: Intravascular laser irradiation of blood
- Control group (Sham Comparator): The steps for the control group are the same as the treatment group, except that the output power is adjusted to zero intensity.
  Interventions: Device: Intravascular laser irradiation of blood (Sham)

INTERVENTIONS:
Device: Intravascular laser irradiation of blood — Low intensity intravascular laser irradiation of blood phototherapy is a method of a 632.8 nm red light penetrate into a vein through fiber and the brightness is 100 fold of the sun. The light accelerates blood and cells circulation in the human body, so that protein molecular structure would promote changes.
  Arms: Treatment group
Device: Intravascular laser irradiation of blood (Sham) — zero intensity of the laser energy
  Arms: Control group

SUMMARY:
This research is designed through randomization, control, and double-blind trial to explore the clinical effectiveness of intravenous laser irradiation of blood for knee degenerative arthritis; and to explore the changes in body's balance function. Furthermore to establish a new way of clinical rehabilitation therapy. The research will further study the special biomarker to investigate the mechanism of low-energy intravenous laser therapy for osteoarthritis.

DETAILED DESCRIPTION:
Background This research is designed through randomization, control, and double-blind trial to explore the clinical effectiveness of intravenous laser irradiation of blood for knee degenerative arthritis; and to explore the changes in body's balance function. Furthermore to establish a new way of clinical rehabilitation therapy. The research will further study the special expression of blood cells after the treatment and as well as the molecular mechanism of low-energy intravenous laser therapy on hematopoietic stem cells. fold of the sun. The light accelerates blood and cells circulation in the human body, so that protein molecular structure would promote changes. Pain control is indicated in such treatment, but still lacking evidence of improving the symptoms of degenerative knee arthritis.

Purpose This research is designed through randomization, control, and double-blind trial to explore the clinical effectiveness of intravenous laser irradiation of blood for knee degenerative arthritis; and to explore the changes in body's balance function. Furthermore to establish a new way of clinical rehabilitation therapy. The research will further study the special biomarker to investigate the mechanism of low-energy intravenous laser therapy for osteoarthritis.

Method The investigators plan to recruit 20 patients who are between the ages of 50 to 75 years old, but younger than 75 years old. The participants are required to have clear conscious and be able to communicate. Their symptoms of degenerative arthritis could be one or both knees which last more than six months; with knee pain greater than 4 points when walking. The treatment group will receive an intravenous helium-neon laser phototherapy. A vein indwelling needle will be placed in their veins located in the upper elbow, and the laser fiber catheter will be introduced through the indwelling cannula. The power is set between 2.5 ~ 3.0Mw, 60 minutes each time, once a day for five consecutive days. The steps for the control group are the same, except that the output power is adjusted to zero intensity. This plan will be explained to the patient in detail during the outpatient visit and patients will sign the consent form upon agreement. Before intravenous laser irradiation, three days, one month, and three months after the therapy, 20 ml of autologous peripheral venous blood need to be drawn for basic blood tests and biomarker tests. At the same time, the clinical functions of patients will be evaluated, including visual analogous scale, Lequesne 's severity index, WOMAC scale, and balance function test.

ELIGIBILITY:
Inclusion Criteria:

* clear conscious and be able to communicate.
* the symptoms of degenerative arthritis could be one or both knees which last more than six months
* with knee pain greater than 4 points when walking

Exclusion Criteria:

* had ever received intraarticular injection with hyaluronic acid or steroid within 6 months
* had ever received nonsteroidal anti-inflammatory drugs or steroid therapy within 1 week
* neoplasm of joint and peripheral soft tissue
* malignancy
* had ever received total knee arthroplasty or other major surgery
* rheumatoid arthritis
* coagulopathy
* unable to take balance test due to other chronic disease

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) of the degree of pain | 3 months
  with the score ranging from 10 (tremendous pain) to 0 (no pain). Measure before intravenous laser irradiation, three days, one month, and three months after the therapy.
The Western Ontario and McMaster Universities Arthritis Index (WOMAC) | 3 months
  Score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. The higher score means more severity. Measure before intravenous laser irradiation, three days, one month, and three months after the therapy.
Lequesne 's severity index | 3 months
  Three domain: pain or discomfort, maximum distance walked, activities of daily living. Score range of 0-26. The higher score means more severity. Measure before intravenous laser irradiation, three days, one month, and three months after the therapy.
Balance function test | 3 months
  Test standing balance,including static, dynamic with opening and closing eyes, and single leg stance. Measure before intravenous laser irradiation, three days, one month, and three months after the therapy.

SECONDARY OUTCOMES:
Serum Interleukin 6 (IL6) | 3 months
  chemiluminescent enzyme immunometric assay method. Measure before intravenous laser irradiation, three days, one month, and three months after the therapy.
Serum cartilage oligomeric matrix protein (COMP) | 3 months
  immunoassay ELISA. Measure before intravenous laser irradiation, three days, one month, and three months after the therapy.
Serum procollagen type II N-terminal propeptide (PIIANP) | 3 months
  ELISA. Measure before intravenous laser irradiation, three days, one month, and three months after the therapy.
Serum calcitonin gene-related peptide (CGRP) | 3 months
  immunosorbent assay (ELISA). Measure before intravenous laser irradiation, three days, one month, and three months after the therapy.
Substance P | 3 months
  Substance P Immunoassay Test. Measure before intravenous laser irradiation, three days, one month, and three months after the therapy.
The number of synovium-derived stem cell with CD73, CD90, CD105 | 3 months
  flow cytometry, Measure before intravenous laser irradiation, three days, one month, and three months after the therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Liang-Cheng Chen, MD,MS, Principal Investigator — Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Locations (1):
- Tri-service general hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang SF, Tsai YA, Wu SB, Wei YH, Tsai PY, Chuang TY. Effects of intravascular laser irradiation of blood in mitochondria dysfunction and oxidative stress in adults with chronic spinal cord injury. Photomed Laser Surg. 2012 Oct;30(10):579-86. doi: 10.1089/pho.2012.3228. Epub 2012 Aug 14. PMID 22891782
- [Background] Thunshelle C, Hamblin MR. Transcranial Low-Level Laser (Light) Therapy for Brain Injury. Photomed Laser Surg. 2016 Dec;34(12):587-598. doi: 10.1089/pho.2015.4051. PMID 28001759
- [Background] de Freitas LF, Hamblin MR. Proposed Mechanisms of Photobiomodulation or Low-Level Light Therapy. IEEE J Sel Top Quantum Electron. 2016 May-Jun;22(3):7000417. doi: 10.1109/JSTQE.2016.2561201. PMID 28070154
- [Background] Munjal A, Bapat S, Hubbard D, Hunter M, Kolhe R, Fulzele S. Advances in Molecular biomarker for early diagnosis of Osteoarthritis. Biomol Concepts. 2019 Aug 9;10(1):111-119. doi: 10.1515/bmc-2019-0014. PMID 31401621
- [Background] Watt FE. Osteoarthritis biomarkers: year in review. Osteoarthritis Cartilage. 2018 Mar;26(3):312-318. doi: 10.1016/j.joca.2017.10.016. Epub 2017 Oct 26. PMID 29107060
- [Background] Campbell DD, Pei M. Surface markers for chondrogenic determination: a highlight of synovium-derived stem cells. Cells. 2012 Nov 16;1(4):1107-20. doi: 10.3390/cells1041107. PMID 24710545